CLINICAL TRIAL: NCT04612556
Title: Efficacy of Mepolizumab in Patients With Late-onset Severe Eosinophilic Asthma and Fixed Obstruction
Brief Title: Efficacy of Mepolizumab in Severe Asthmatics on a Long Term (MESILICO)
Acronym: MESILICO
Status: Active, not recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: NHS Pulmonary Clinic G. Papanikolaou Hospital, Thessaloniki, Greece (Unknown); Pulmonary Clinic of Army Hospital Thessaloniki Greece (Unknown); Pulmonary Clinic, Democritus University of Thrace (Unknown); Pulmonary Clinic, University of Ioannina (Unknown); 1st Pulmonary Clinic, Kapodistrian University of Athens (Unknown); 2nd Pulmonary Clinic, Kapodistrian University of Athens (Unknown); NHS 7th Pulmonary Clinic, Sotiria Hospital, Athens (Unknown)
Responsible Party: Principal Investigator, Associate Prof Konstantinos Porpodis, Assistant Professor of Pulmonology, Aristotle University Of Thessaloniki
Other Study IDs: Study 12316
Record Dates: First submitted 2020-09-18; First posted 2020-11-03 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Eosinophilic; Severe Asthma; Late-Onset Asthma
Keywords: severe eosinophilic asthma, late-onset, fixed obstruction
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — mepolizumab; Biological Products; Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood, bronchial washing, sputum and sputum supernatant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- late-onset severe eosinophilic asthma and fixed obstruction: Patients with late-onset severe eosinophilic asthma and fixed obstruction will be administered Mepolizumab (100 MG), subcutaneusly every 30 days
  Interventions: Drug: Mepolizumab 100 MG [Nucala]

INTERVENTIONS:
Drug: Mepolizumab 100 MG [Nucala] — subcutaneous injection once a month
  Other Names: biological/vaccine

SUMMARY:
Interleukin (IL)-5 is the main cytokine responsible for the activation of eosinophils, hence therapeutic strategies have been investigated and developed for clinical use. Biologics targeting IL-5 and its receptor (first mepolizumab and subsequently, reslizumab and benralizumab), have been recently approved and used as add-on therapy for severe eosinophilic asthma resulting in a reduction in the circulating eosinophil count, improvement in lung function and exacerbation reduction in patients with severe asthma.

Response to biologic therapies in severe asthma is variable, with patients being either non-responders, responders or super-responders. There is currently no explanation for this broad variation in response. It is important to examine whether these patients have distinct characteristics that could help the treating physician in making the correct diagnosis in clinical practice.

Aim of this clinical study is to evaluate the efficacy of mepolizumab, a humanized IL-5 antagonist monoclonal antibody in patients with late-onset severe eosinophilic asthma with fixed obstruction and to identify the characteristics of non-responders and super-responders under mepolizumab treatment. This study is considered as non-interventional and every procedure included is happening in a clinical routine for the diagnosis and phenotyping of the asthmatic patients.

Hypothesis includes the efficacy of mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction and relation to clinical and inflammatory biomarkers.

Patients will be collected from the outpatient clinics of bronchial asthma from each site included (8 in number) which cover the whole population of Greece.

Overall, this is a prospective multicenter study including eight Pulmonary Clinics. Five Pulmonary University Clinics, two of National Health System and one Army General Hospital in Thessaloniki. The study will include a screening period of up to 2 weeks to assess eligibility and obtain written informed consent, a mepolizumab treatment period of 52 weeks, once every 4 weeks, including follow up visits every 3 months during treatment. The study population will consist of 45 patients with late-onset severe eosinophilic asthma and fixed obstruction receiving mepolizumab, aged 20 and above.

DETAILED DESCRIPTION:
Scientific rationale Interleukin (IL)-5 is the main cytokine responsible for the activation of eosinophils, hence therapeutic strategies have been investigated and developed for clinical use. Biologics targeting IL-5 and its receptor (first mepolizumab and subsequently, reslizumab and benralizumab), have been recently approved and used as add-on therapy for severe eosinophilic asthma resulting in a reduction in the circulating eosinophil count, improvement in lung function and exacerbation reduction in patients with severe asthma.

Response to biologic therapies in severe asthma is variable, with patients being either non-responders, responders or super-responders. There is currently no explanation for this broad variation in response. It is important to examine whether these patients have distinct characteristics that could help the treating physician in making the correct diagnosis in clinical practice.

Aim of this clinical study is to evaluate the efficacy of mepolizumab, a humanized IL-5 antagonist monoclonal antibody in patients with late-onset severe eosinophilic asthma with fixed obstruction and to identify the characteristics of non-responders and super-responders under mepolizumab treatment. This study is considered as non-interventional and every procedure included is happening in a clinical routine for the diagnosis and phenotyping of the asthmatic patients.

Several methods are used to investigate airway inflammation: direct measurements (like bronchial biopsies or bronchoalveolar lavages) and indirect methods (like symptom assessment, blood sample analysis and lung function tests). The direct techniques have the advantage of reliably assessing the airway inflammation, but they are invasive and not feasible at large scale because of patient discomfort and the risk incurred. As for the indirect methods, they poorly correlate with the direct assessment of airway inflammation.

In this study, among patients' clinical characteristics spirometry, biomarkers of inflammation (blood eosinophils, FeNO, IgE levels), impulse oscillometry (IOS) and the thickening of basement membrane via bronchoscopy will be evaluated. It is suggested that late-onset severe eosinophilic asthmatic patients with fixed obstruction who do not respond to the usual treatment (ICS/LABA/LAMA) appear with increased smooth muscle mass. However, the precise effects of increased airway smooth muscle mass on airway narrowing are not known and may vary with disease severity. In addition, biomarkers of inflammation will also be evaluated before and after 52-week mepolizumab treatment in biological fluids (serum, sputum, sputum supernatant and bronchial samples). Biomarkers of inflammation are very important to identify responders to non-responders.

More specific, IOS has been introduced as an alternative technique to assess lung function with particular application to asthma. This technique is noninvasive, easily performed during tidal breathing and requires only minimal patient cooperation.

Sputum collection is another way to sample cells from the airways and allows the direct assessment of airway inflammation. Furthermore, examples with sputum supernatant include the analysis of mediators and the assessment of the chemotactic activity of the sample for eosinophils. The sputum cells can also be analyzed by flow cytometry which allows, among others, immunophenotyping and sorting cells. Furthermore, sputum cells can be cultured, and their mediator production can be measured in vitro. It is worth noting that in this case, the mediator content is different from what can be found in sputum supernatant. Indeed, mediators in sputum supernatant may be influenced by secretions from airway resident cells and by plasma exudation, contrary to the sputum cell culture model. Finally, immunocytochemistry and in situ hybridization can also be performed using sputum cells.

Although phenotypes, blood eosinophils, and serum IgE levels have been proposed for use as a reference, there is a dissociation between the blood immune-cell level and the airway epithelium immune reaction, as confirmed in previous studies. Airway epithelium immunohistochemistry staining for targeted immune cells has been used to determine various types of airway inflammation; however, this technique is rarely used in a clinical setting. Previous studies have revealed the relative safety of performing bronchoscopy biopsies for patients with severe asthma. Among the sampling techniques used for tissue diagnosis, including nasal biopsies, nasal or bronchial brushing, and bronchoalveolar lavage, bronchoscopy-guided bronchial epithelium sampling provides more accurate information about the epithelial and inflammatory cells in the tissue context. It is thus a powerful tool for selecting the most suitable biologics in difficult clinical conditions.

Besides, asthmatic disease is characterized by a chronic mucosal inflammatory process, which results in irreversible changes of the bronchial wall, known today as "bronchial remodeling". Glandular and smooth muscle fibers hyperplasia and/or hypertrophy, goblet cells hyperplasia, and variable thickening of basement membrane (BM) present under the respiratory epithelium are part of these morphological changes. the changes generated at the epithelium-connective interface account for an "adaptive response" to inflammatory stress and sporadic bronchoconstriction. However, current data on BM reactivity in asthmatic patient are still incomplete for an accurate assessment of its involvement in pathogenesis and specifically in bronchial wall remodeling, mainly as collagen deposits in lamina reticularis are not correlated to the degree of disease severity.

Moreover, it is increasingly evident that severe asthma is not a single disease, as evidenced by the variety of clinical presentations, physiologic characteristics, and outcomes seen in patients with asthma. To better understand this heterogeneity, the concept of asthma phenotyping and endotyping has emerged. Phenotyping integrates both biological and clinical features, from molecular, cellular, morphologic, and functional to patient-oriented characteristics with the goal to improve therapy. Ultimately, these phenotypes evolve into asthma "endotypes," which combine clinical characteristics with identifiable mechanistic pathways. Biomarkers, defined as characteristics that can be objectively measured and serve as an indicator of underlying biological processes or pathogenesis, are crucial in defining phenotypes and endotypes. In asthma, genetic polymorphisms, measures of airway physiology, and levels of inflammatory mediators in urine, blood, sputum, tissue, exhaled gas, and breath condensate have all been studied as potential markers to improve and objectify asthma diagnosis and management. Developing such tools will allow us to phenotype and endotype the various clinical patterns described in asthma, with the ultimate goal of tailoring therapy based on a specific biomarker profile. Biomarkers can then be used to help better understand the pharmacologic response to an intervention and adjust therapy accordingly.

Biomarkers have been critical for studies of disease pathogenesis and the development of new therapies in severe asthma. In particular, biomarkers of type 2 inflammation have proven valuable for endotyping and targeting new biological agents. Because of these successes in understanding and marking type 2 inflammation, lack of knowledge regarding non-type 2 inflammatory mechanisms in asthma will soon be the major obstacle to the development of new treatments and management strategies in severe asthma. Other potential biomarkers include innate lymphoid cells, IL-33 or thymic stromal lymphopoietin.

Recent publications confirmed crucial regulatory role of miRNAs in the pathomechanism of asthma. Some single miRNAs or their sets hold the promise for their use as asthma biomarkers facilitating diagnosis or prediction of treatment outcomes. They are also possible target of future therapies. The studies in this field are lacking though. Recently it has been shown that most of the involved miRNAs increase secretion of Th2 cytokines, decrease secretion of Th1 cytokines, promote differentiation of T cells towards Th2 or play a role in hyperplasia and hypertrophy of bronchial smooth muscle cells. The profiles of miRNAs correlate with clinical characteristics, including lung function, phenotype and severity of asthma.

Most industry sponsored biologic clinical trials have effectively used the above approach by selecting study subjects that resemble the severe asthma clinical phenotypes of SARP (high-intensity controller medication regimens, frequent exacerbations, and low lung function), but then require an elevated biomarker (in blood, exhaled gas, or sputum) that should identify patients most likely to be responders to a specific immunomodulator within those clinical phenotypes. The biologics in recently published clinical trials target type 2 inflammatory pathways and restrict participation to subjects with elevated type 2 biomarkers (blood or sputum eosinophils or FeNO). Post hoc responder analyses to "group" biomarkers to better understand which patients have the greatest benefit from a biologic immunomodulator will lead to an understanding that concurrent elevations in more than 1 type 2 inflammatory biomarker may further identify "high responder" patients.

Hypothesis includes the efficacy of mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction and relation to clinical and inflammatory biomarkers.

Research questions Is there any improvement in exacerbation rate in late-onset severe eosinophilic asthmatic patients under mepolizumab treatment during their 1st year of treatment and what are the characteristics of non-responders and super-responders? Is there any improvement in smooth muscle cells remodeling? Are there any biomarkers to predict response to mepolizumab treatment in late-onset severe eosinophilic asthmatic patients? Is there any improvement in respiratory parameters? Is there any improvement in asthma control and patients' quality of life? Objectives

The primary objectives of this study are:

1. To demonstrate the effect of mepolizumab treatment in exacerbation rate in late-onset severe eosinophilic asthmatic patients with fixed obstruction.
2. To identify characteristics of non-responders and super-responders.
3. Stydy's extension to identify any improvement in airway remodeling after 156 months of treatment

The key secondary objectives of this study are:

1. Any improvement in remodeling (thickening of bronchial smooth muscle cells).
2. Any possible biomarkers of response.
3. Any improvement in respiratory parameters in asthma control and in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction.

Study design and Methods Patients will be collected from the outpatient clinics of bronchial asthma from each site (8 in number) which cover the population of Greece. All these Clinics are included to reinforce the recruitment as well as to include bronchoscopist experts with international impact. Due to the current situation concerning Covid-19 pandemic, the investigators assume that this clinical study does not interfere with the workload in our Clinics.

Overall, this is a prospective multicenter study including eight Pulmonary Clinics. Five Pulmonary University Clinics, two of National Health System and one Army General Hospital.

The study will include a screening period of up to 2 weeks to assess eligibility and obtain written informed consent, a mepolizumab treatment period of 52 weeks, once every 4 weeks, including follow up visits every 3 months during treatment.

The extension of the protocol includes a treatment period of 156 weeks of treatment.

The study population will consist of 45 patients with late-onset severe eosinophilic asthma and fixed obstruction receiving mepolizumab aged 20 and above.

Study participation, assessment and follow up:

Screening: Investigators will screen selected subjects to the participated clinics (Severe Asthma outpatient clinics). Subjects will come in to sign consent. Clinical assessment and procedures and structural interviews will be performed during screening. Subjects that are eligible/able to complete the screening Visit may do so, on the same day, and if necessary, they will complete their baseline assessment within 2 weeks. Subjects with an ongoing asthma exacerbation should have their screening and treatment initiation visit delayed until the investigator considers the subject has returned to their baseline asthma status. If the 2-week screening period has elapsed then the subject should be considered a screening failure. Subjects will remain on their current maintenance therapy throughout screening periods. Eligibility of the patients will be based on the criteria listed in the next sections.

Asthma exacerbation history for the last 12 months will be reported at screening visit. Also, exacerbations will be evaluated at each visit as reported.

Vital signs will be performed at screening visit, at baseline and every 3 months. Measurements will include systolic and diastolic blood pressure, pulse rate and body temperature.

Height in centimeters (cm) and body weight in kilograms (kg) will be measured at screening visits. Body Mass Index (BMI) will be calculated as the weight in kg divided by the height in meters squared

Laboratory evaluation (Hematology, Blood chemistry, Urinalysis):

Venous blood and urine will be collected at baseline. Hematology: Hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, and platelet will be measured in the laboratory of each site's hospital. Basic clinical chemistry and urinalysis will be evaluated. Collection of urine for female subjects will also evaluate pregnancy.

IgE levels will be evaluated at screening visit using immunoCAP tests and will be reported as IU/mL.

The following Questionnaires will be administered: 1) the Asthma Control Questionnaire (ACQ-5) and Asthma Control Test (ACT) to assess current asthma control; 2) the Asthma Quality of Life Questionnaire (AQLQ+12) to assess quality of life and psychological morbidity. To further asses sleeping quality 1) Athens Insomnia Scale (AIS), 2) Epworth Sleepiness Scale (ESS), 3) St. George's Respiratory Questionnaire (SGRQ) and 4) WHO (Five) Well-Being Index (WHO-5), 5) Fatigue Severity Scale (FSS).

Exhaled nitric oxide (NO) will be measured at baseline and every 3 months according to the American Thoracic Society Guidelines and as specified by the manufacturer. FeNO levels will be reported as parts per billion. Measurements will be made before spirometry is performed.

Venous blood samples will be retrieved between 8 to 10 am, at baseline and every 3 months during the 52-week period with mepolizumab treatment. Absolute blood eosinophil count will be reported as cells/μl.

Spirometry: Spirometry A will be conducted, using the site's own equipment at the visits (baseline and every 3 months). All clinic visits must occur in the morning. During the treatment period the spirometry will meet the current ATS/ERS guidelines and the spirometer must produce a printout of all data generated, which should be stored in the subject's notes. The spirometer will be calibrated in accordance with the manufacturer's instructions. Spirometry must be performed at the same time (±1 hour) of the Visit 0 spirometry. Subjects should try to withhold short-acting beta-2-agonists (SABAs) for ≥4 hours and LABAs for ≥15 hours prior to clinic visit, if possible (GINA 2019). Assessments to be recorded will include FEV1, FVC, FEV1/FVC%, PEF and FEF25-75. Post-bronchodilator measurements will be taken at every visit, using 200-400mcg albuterol or equivalent.

Spirometry B will be conducted, using the site's own equipment at the visits (baseline, after 6 months and after treatment at 52 weeks timepoint). Spirometry B includes diffusion, pulmonary volumes and capacities.

Impulse oscillometry (optional):

Impulse Osillometry (IOS) will be conducted at baseline and after 52 weeks of treatment. IOS includes resistance at 5 Hz-resistance at 20 Hz (R5-R20), a measure reflecting respiratory resistance of small to midsized conductive and peripheral airways, AX, a measure reflecting distensibility of the peripheral lungs (namely the parenchyma and small peripheral airways), and the respiratory system reactance (X5), a measure reflecting inertance and elasticity or capacitance (including small peripheral airways).

Therapy with biologics:

Upon completion of the screening visits the participant may initiate treatment with biologic therapy (mepolizumab) within a month. During therapy subjects will be under the care of the pulmonologist who had referred them to the research group for taking part into the study. These pulmonologists will be termed as 'associate pulmonologists. Treatment will be provided as per product manufacturer instructions.

Associate pulmonologists providing biologic treatment during the study will require to sign an agreement to conduct the study in compliance with the protocol, to acknowledge that he/she is responsible for medical conduct and for study conduct, and to ensure that the associate (and their colleagues and employees) assisting in the conduct of the study are informed about their obligations. Mechanisms will be in place to ensure that associate staff receives the appropriate information and support by the research group throughout the study.

Follow up during biologic therapy: At initiation and at every visit for biologic therapy administration collection of information will be performed by the associate pulmonologist, and with support by the research group if requested by the associate pulmonologist e.g., researchers via telephone or face-to-face contact will interview the patient. Furthermore, compliance will be recorded form the physician based on patient's oral confirmation. Date form of drug administration will be recorded at every visit, as well as immediate and delayed adverse effects.

Safety monitoring:

Recorded adverse events (AEs) will be monitored and collated as required in study reports. An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study entry. Medical conditions/diseases present before starting study drug are only considered adverse events if they worsen after starting study drug. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy. Also, adverse events related to Covid-19 are included. If a partner pulmonologist or research staff becomes aware of an AE associated with a product, it can be reported to the manufacturer according to their local standard practice for spontaneous AE reporting. A copy of the report should also be sent to the study coordinator. Serious adverse events (SAE) will be reported in the eCRF pages and within 24 hours all the investigators will have the responsibility to inform the Central Committee in Thessaloniki. Then the Central Committee will inform the scientific board and the Greek Medical Agency. Also, medical and scientific judgment will be exercised by the principal investigator of each center with the Central Committee, in deciding whether the subject should stop the treatment or not.

Pregnancy report:

Initially, female patients at screening will have to do a pregnancy test. During treatment, if a female subject reports a pregnancy to us, she will be asked to withdraw from the study (to prevent bias) Then, she will be asked if she would like to keep getting the treatment outside of this protocol and be monitored at each center's outpatient clinic.

Pre-screening and Screening Failures:

Subjects will be assigned a study number at the time of signing the consent. Subjects who signed but do not progress to the screening visits assessment will be deemed a pre-screen failure. No data will be captured in the database for these subjects.

Subjects that complete at least one of the two screening visits, but do not initiate biologic therapy will be designated as screening failures. Information to be collected for pre-screening and screening failures will be detailed in the database completion.

Withdrawal Visit:

If a participant decides to withdraw from the study during follow-up (for any reason other than loss to follow up), they may be asked to attend a withdrawal visit (if deemed necessary by investigator and subject to consent). During the visit, the participant may be asked questions about their current conditions as part of clinical information collection such as: asthma and nasal symptoms, exacerbations and the progression of treatment being received.

Blood samples' collection and processing:

Blood samples will be collected at baseline visit, at 6 months and after treatment completion. After collecting the blood samples, they will be left undisturbed for about half an hour for complete clot formation. The sample will then be centrifuged to separate the serum from the clot. After centrifugation the serum will be stored at -20° C in eppendorf tubes till the analysis was done. Blood phenotyping will also be evaluated by flow cytometry.

Induced sputum (optional):

Induced sputum will be performed at baseline before treatment initiation and after completion of treatment according to the ERS Task Force report where a detailed expert consensus-based recommendation for induced sputum processing is suggested.

At the visits, sputum induction will be performed after the routine spirometric assessments have been completed.

The induced sputum will be processed within two hours of the end of the induction procedure at the research site. Sputum cells and cell suspension supernatant will be stored at -80ºC for analysis. After collecting the induced sputum, the supernatant of the sample will be stored at -20° C in eppendorf tubes till the analysis was done. Following these procedures, laboratory evaluation of the sputum is next according to guidelines.

Bronchoscopy, bronchial biopsies and washing samples' collection and processing (optional): At the visits, endoscopy with bronchial biopsies, bronchial washing sample (Visit 0b) will be performed upon patient's written consent. In specific, a separate inform consent will be included to be signed from each patient. Bronchoscopy will be performed at two time-points (baseline before treatment initiation and after the completion of treatment). Flexible bronchoscopy and diagnostic techniques were performed under monitored anesthesia care as recommended by the American Thoracic Society and the British Thoracic Society.

Tissue samples will be fixed in inflation or immersion using formaldehyde or glutaraldehyde and embedded in paraffin. Airways will be systematically sampled or obtained during diagnostic dissection at the discretion of the pathologist. Consecutive sections of 0.5, 5 and 30 μm thickness were cut from each block and stained using the Masson's trichrome technique, haematoxylin and eosin, and haematoxylin, respectively. Immunohistochemical staining will be done done with the following mAbs: anti-mast cell tryptase clone AA1 (Dako UK), anti-alpha smooth muscle actin clone 1A4 (Dako UK), anti-eosinophil major basic protein clone BMK-13 (Monosan, Netherlands), anti-neutrophil elastase clone NP57 (Dako UK), and anti-endothelium clone EN4 (Monosan, Netherlands) or appropriate isotype controls were used.

The endobronchial biopsies will be assessed by a single observer blinded to the clinical characteristics (ZEN 2012 image analysis software for light microscopy, Carl Zeiss AG, Germany) and will be expressed as the mean of measurements undertaken from a minimum of two sections either from independent biopsies or as non-contiguous tissue sections at least 20μm apart from the same biopsy. Epithelial integrity will be assessed by measuring the lengths of intact and denuded epithelium. These will be expressed as percentage of all the reticular basement membrane (RBM) length. Vascularity will be measured using the Chalkley count, a surrogate of both vessel density and vascular area. A Chalkley eyepiece graticule (NG52 Chalkley Point Array, Pyser-SGI Ltd, UK) will be used at x200 to measure Chalkley counts in four non-overlapping vascular hotspots (6). Airway smooth muscle content will be determined as the proportion of the total area. Inflammatory cells were expressed as the number of nucleated cells/area of lamina propria.

Bronchial washing samples will be immediately transported to the laboratory, to be stored at -80 degrees. Examination of bronchial washing fluids will be performed at a later stage to determine several biomarkers.

Analysis of biomarkers of inflammation with Flow Cytometry Analysis (FACS) or ELIZA:

Biomarkers included before and after treatment with mepolizumab in two or three timepoints, (at baseline, at 6 months treatment and after treatment completion visit): lymphocyte subsets, Th2/Th17 cytokines, chemokines, microRNAs expression to be quantitated by flow cytometry or ELISA) in biological fluids (blood, serum, bronchial washing, sputum and sputum supernatant).

Panel kits and appropriate antibodies will be tested by Flow Cytometer Analysis using a BD FACS Calibur system (BD Biosciences, San Jose, CA), according to the manufacturer's recommendations and instructions.

ELISA (enzyme-linked immunosorbent assay) is a plate-based assay technique designed for detecting and quantifying substances such as peptides, proteins, antibodies and hormones. ELISA kits will be analyzed using VICTOR X3 spectrophotometer according to the manufacturer's recommendations and instructions.

Allergy testing (If applicable) The patients' atopic status will be evaluated (if not available) at screening visit by the skin prick test (SPT) to a standard panel of aeroallergens for detecting total IgE antibodies against various common inhalant allergens.

Database An electronic data collection platform will be the method used at baseline every 3 months until 1 year follow up for this database. During treatment visits paper forms/questionnaires will be completed by the associate pulmonologist. Each site will entry specific data in an electronic database. Each patient is uniquely identified by a Subject number which is composed by the site number assigned by the responsible monitoring site and a sequential number assigned by the investigator. Upon signing the informed consent form, the patient is assigned the next sequential number by the investigator. The site must contact the central research personnel and provide the requested identifying information for the patient as registered into the electronic database. The treatment visit forms will also be sent to the central research personnel. The authorized study personnel will be responsible for data collection, editing, and also protecting the data being collected at their own site and the database is backed up on a daily basis. Quality review/control will be the joint responsibility of all individuals involved and the central research personnel [data custodian].

Sample size calculation G power analysis Sample size is calculated using the G*Power software (Die Heinrich-Heine-Universität Düsseldorf, Germany). The difference in annual exacerbation rate of the patients with late onset severe eosinophilic asthmatics before and after Mepolizumab treatment with is the primary endpoint of the study. In the DREAM study (one of the only two studies that has reported results similar to our primary endpoint so far) it was reported that the annual exacerbation rate of patients with severe Asthma declined from 3.6 to 1.33 after the initiation of treatment with Mepolizumab. Using this data and a two-sided test, with a power at 0.95 and a level of statistical significance at 0.05, the investigators calculated an effect size of 0.556, which indicated a total sample size of 45 participants.

Statistical Plan Analysis Statistical analysis will be performed using the SPSS (version 21.0 IBM SPSS statistical software, Armonk, NY, USA). Categorical variables will be stated as numbers (n) and percentages (%), continuous variables as mean ± SD if normally distributed, or median and interquartile ranges if otherwise. Where necessary variables without a normal distribution will be transformed. P < 0.05 was accepted as statistically significant. Shapiro-Wilk test will be performed in order to separate parametric from non-parametric variables. Paired-Samples T Test for parametric or Wilcoxon Signed Ranks test for non-parametric variables will be used to detect differences in the variables measured before and after Mepolizumab treatment.

There is no comparator arm as every patient is control to himself. There are baseline characteristics (clinical and laboratory biomarkers) that are going to be measured at baseline, every 3 months and after 52-week treatment completion. Study endpoints include the analysis of all those biomarkers as the identification of the characteristics of non-responders and super-responders. Also, secondary endpoints include the evaluation of the biomarkers mentioned in the methods as assessments. Statistical analysis will be performed initially with the number of patients that have completed the 52-week period of treatment. Secondly, patients that have not completed the 52-week treatment will be analyzed separately and finally these two groups are going to be compared to each other.

More specifically, with univariate analysis (two-sided independent sample tests) the investigators will test for associations/correlations between all baseline outcomes compared with the ones after mepolizumab treatments (every 3 months until 1 year of treatment): biomarkers in sputum and in blood, clinical outcomes. Similarly, univariate associations between outcomes and personal/demographic characteristics will be tested for identifying potential confounders. Significant associations will be then tested with adjusted regression models. Associations/correlations will be evaluated separately at baseline clinical characteristics and every 3 months follow up during treatment as well as at baseline and after 1 year of mepolizumab treatment. Besides, subgrouping analysis will be performed for each biomarker for the identification of biomarker level to treatment response.

Paired-Samples T Test for parametric or Wilcoxon Signed Ranks test for non-parametric variables will be used to detect differences in the variables measured before and after Mepolizumab treatment. In specific, levels of biomarkers at baseline will be compared to levels after 1-year of mepolizumab treatment.

Overall response to treatment in one year (from baseline to 1-year post treatment initiation) for each outcome will be measured with paired test of dependent samples (parametric and non-parametric paired tests) in each patient. Then response to treatment will be defined as the change (absolute and % change) of the outcome in one year. The investigators will assess predictors influencing response to treatment (change) such as biomarkers by using multiple regression models for each clinicopathological outcome. For outcomes with more than 2 observations per subject during the study period the investigators will use mixed models using the repeated measurements of the outcome. All tests will be 2-sided with a statistical significance level at 5%.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria

* Written informed consent must be obtained at screening visit, before any assessment will be performed. Subjects should be able to provide informed written consent (study participation informed consent form): Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Confirmed asthma diagnosis and severity and treatment requirements.
* Fixed airway obstruction (FAO) where post-bronchodilator treatment ratio of forced expiratory volume in 1 second [FEV1] to forced vital capacity [FVC] is below < 70%.
* Confirmed optimized management skills (inhaler technique, education, adherence)
* Triggers and relevant co-morbidity have been assessed and managed Triggers such as smoking, beta-blockers, aspirin/NSAIDs, allergen exposure; Comorbidities such as rhinitis, obesity, GERD, OSA, VCD, depression/anxiety.
* Severe asthmatics with blood eosinophils ≥150cells/ul at screening visit or ≥300cells/ul the last 12 months.
* Patients with late-onset severe according to ERS/ATS guidelines eosinophilic asthma and fixed obstruction under the treatment of high dose of ICS+LABA±LAMA (late-onset asthma determined as age at diagnosis from 20 years and above)
* Patients with late-onset severe eosinophilic asthma with history ≥ 1 exacerbation the previous year under the treatment of high dose of ICS+LABA±LAMA.
* Asthma Exacerbation: Subjects with an ongoing asthma exacerbation should have their screening and treatment initiation visit delayed until the investigator considers the subject has returned to their baseline asthma status. If the 4-week screening period has elapsed then the subject should be considered a screening failure. An exacerbation is defined as worsening of asthma requiring the use of systemic corticosteroids and/or emergency department visit, or hospitalization. For subjects on maintenance oral corticosteroids, an exacerbation requiring oral corticosteroids was defined as the use of oral/systemic corticosteroids at least double the existing dose for at least 3 days.
* Maintenance Asthma Therapy: No changes in the dose or regimen of baseline ICS and/or additional controller medication during the screening period (except for treatment of an exacerbation).
* Meet requirements for biologic therapy with mepolizumab.

Exclusion Criteria:

* Asthma exacerbation, within 6 weeks prior to screening that required hospitalization or emergency room visit.
* Prior use of other biologics (including but not limited to Omalizumab, Reslizumab, Dupilumab, Benralizumab etc., for asthma or any other indications) that has potential to interfere/ affect disease progression, in the previous 6 months.
* Pregnant or nursing women, or women of child-bearing potential.
* History of malignancy of any organ system or any other serious co-morbidities defined by the treating physician.
* Patients with a history of conditions other than asthma that could result in elevated eosinophils (e.g. hypereosinophilic syndromes, Churg-Strauss Syndrome, eosinophilic esophagitis).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 45 patients with late-onset severe eosinophilic asthma and fixed obstruction receiving mepolizumab aged 20 and above.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in exacerbation rate | through study completion, 156 weeks
  Mesurement of the change in exacerbation rate in each late-onset severe eosinophilic asthmatic patient with fixed obstruction under mepolizumab treatment for 52 weeks of treatment.
Identification of clinical characteristics of response, change in Forced Expiratory Volume (FEV1) | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  FEV1 change from baseline, before treatment initiation, compared to measurements every 3 months until 1 year of treatment. FEV1 is the maximal amount of air you can forcefully exhale in one second measured by spirometry.
Identification of clinical characteristics of response, change in blood eosinophil levels. | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  Change from baseline, before treatment initiation, compared to measurements every 3 months until 1 year of treatment.
Identification of clinical characteristics of response, change in FENO levels. | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  Change from baseline, before treatment initiation, compared to measurements every 3 months until 1 year of treatment.
Identification of clinical characteristics of response, change in Asthma Control Questionnaire | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: the Asthma Control Questionnaire (ACQ-5) to assess current asthma control.
  Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
Identification of clinical characteristics of response, change in Asthma Control Test | through study completion,156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: Asthma Control Test (ACT) to assess current asthma control.
  The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Identification of clinical characteristics of response, change in Asthma Quality of Life Questionnaire | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: the Asthma Quality of Life Questionnaire (AQLQ+12) to assess quality of life and psychological morbidity.
  Scores range 1-7, with higher scores indicating better quality of life.
Identification of clinical characteristics of response, change in Athens Insomnia Scale | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: Athens Insomnia Scale (AIS) to assess sleeping quality.
  Total score range form 0 to 24 with higher scores indicating worst sleeping quality. AIS includes 8 questions with scores range from 0 (meaning that the item in question has not been a problem) to 3 (indicating more acute sleep difﬁculties).
Identification of clinical characteristics of response, change in Epworth Sleepiness Scale | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: Epworth Sleepiness Scale (ESS) to assess sleeping quality.
  The total score can range from 0 to 24. Higher scores indicate increased sleepiness.
Identification of clinical characteristics of response, change in St. George's Respiratory Questionnaire | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: St. George's Respiratory Questionnaire (SGRQ) to assess sleeping quality.
  Scores range from 0 to 100, with higher scores indicating more limitations.
Identification of clinical characteristics of response, change in WHO (Five) Well-Being Index | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: WHO (Five) Well-Being Index (WHO-5) to assess sleeping quality.
  The total raw score ranges from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Identification of clinical characteristics of response, change in Fatigue Severity Scale | through study completion, 156 weeks
  Identification of any improvement in patients' quality of life during mepolizumab treatment in late-onset severe eosinophilic asthmatic patients with fixed obstruction, from baseline, before treatment initiation, compared to every 3 months until 1 year of treatment. Questionnaire included: Fatigue Severity Scale (FSS) to assess sleeping quality.
  FSS includes a 9-item questionnaire with questions scored on a 7 point scale with 1 meaning strongly disagree and 7 meaning strongly agree. Scores range from 9 to 63. Higher the score indicates greater fatigue severity.
Change in smooth muscle cell mass | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders
Change in Basement Membrane Thickness | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders

SECONDARY OUTCOMES:
Change in smooth muscle cell mass | through study completion, 156 weeks
  The identification of clinical characteristics of non-responders and super-responders.
  Any improvement in smooth muscle cell mass will be measured as change from baseline compared to measurement after 1 year of treatment.
  Increased smooth muscle cell mass indicates airway remodeling and loss of pulmonary function.
  Smooth muscle cell mass will be determined through the epithelial integrity, reticular basement membrane length and vascularity area.
Change of T-lympocytes percentages | through study completion, 156 weeks
  To identify any possible biomarkers of response of non-responders versus super-responders in different biological fluids as peripheral blood, bronchial washing, sputum, sputum supernatant.
  The identification of clinical characteristics of non-responders and super-responders.
  Change from baseline compared to measurements after 6 months and after 1 year of mepolizumab treatment.
Change of cytokine and protein levels | through study completion, 156 weeks
  To identify any possible biomarkers of response of non-responders versus super-responders in different biological fluids as peripheral blood, bronchial washing, sputum, sputum supernatant.
  The identification of clinical characteristics of non-responders and super-responders.
  Change from baseline compared to measurements after 6 months and after 1 year of mepolizumab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Porpodis, Assist Prof, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Pulmonary Clinic of Aristotle University of Thessaloniki, George Papanikolaou Hospital, Thessaloniki, Exochi, Greece

IPD SHARING:
Plan to Share IPD: Yes
The results have not yet been published in a peer-reviewed journal. A reference of the published article will be shared here.
Supporting Information: Study Protocol, CSR
Time Frame: Starting 9 months after publication and ending 36 months following article publication.
Access Criteria: Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis, data will be shared. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
  Information regarding submitting proposals and accessing data may be found at (Link to be provided).

REFERENCES:
- [Background] Goldstein RA, Rohatgi PK, Bergofsky EH, Block ER, Daniele RP, Dantzker DR, Davis GS, Hunninghake GW, King TE Jr, Metzger WJ, et al. Clinical role of bronchoalveolar lavage in adults with pulmonary disease. Am Rev Respir Dis. 1990 Aug;142(2):481-6. doi: 10.1164/ajrccm/142.2.481. PMID 2200319
- [Background] Carr TF, Zeki AA, Kraft M. Eosinophilic and Noneosinophilic Asthma. Am J Respir Crit Care Med. 2018 Jan 1;197(1):22-37. doi: 10.1164/rccm.201611-2232PP. No abstract available. PMID 28910134
- [Background] Efthimiadis A, Spanevello A, Hamid Q, Kelly MM, Linden M, Louis R, Pizzichini MM, Pizzichini E, Ronchi C, Van Overvel F, Djukanovic R. Methods of sputum processing for cell counts, immunocytochemistry and in situ hybridisation. Eur Respir J Suppl. 2002 Sep;37:19s-23s. doi: 10.1183/09031936.02.00001902. No abstract available. PMID 12361358
- [Background] Bara I, Ozier A, Tunon de Lara JM, Marthan R, Berger P. Pathophysiology of bronchial smooth muscle remodelling in asthma. Eur Respir J. 2010 Nov;36(5):1174-84. doi: 10.1183/09031936.00019810. PMID 21037369
- [Background] Rasmussen F, Taylor DR, Flannery EM, Cowan JO, Greene JM, Herbison GP, Sears MR. Risk factors for airway remodeling in asthma manifested by a low postbronchodilator FEV1/vital capacity ratio: a longitudinal population study from childhood to adulthood. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1480-8. doi: 10.1164/rccm.2108009. PMID 12045120
- [Background] Fitzpatrick AM, Moore WC. Severe Asthma Phenotypes - How Should They Guide Evaluation and Treatment? J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):901-908. doi: 10.1016/j.jaip.2017.05.015. PMID 28689840
- [Background] Maneechotesuwan K. Role of microRNA in severe asthma. Respir Investig. 2019 Jan;57(1):9-19. doi: 10.1016/j.resinv.2018.10.005. Epub 2018 Nov 16. PMID 30455067
- [Background] Yancey SW, Keene ON, Albers FC, Ortega H, Bates S, Bleecker ER, Pavord I. Biomarkers for severe eosinophilic asthma. J Allergy Clin Immunol. 2017 Dec;140(6):1509-1518. doi: 10.1016/j.jaci.2017.10.005. PMID 29221581
- [Result] Albers FC, Papi A, Taille C, Bratton DJ, Bradford ES, Yancey SW, Kwon N. Mepolizumab reduces exacerbations in patients with severe eosinophilic asthma, irrespective of body weight/body mass index: meta-analysis of MENSA and MUSCA. Respir Res. 2019 Jul 30;20(1):169. doi: 10.1186/s12931-019-1134-7. PMID 31362741
- [Result] Bennett GH, Carpenter L, Hao W, Song P, Steinberg J, Baptist AP. Risk factors and clinical outcomes associated with fixed airflow obstruction in older adults with asthma. Ann Allergy Asthma Immunol. 2018 Feb;120(2):164-168.e1. doi: 10.1016/j.anai.2017.10.004. Epub 2017 Dec 28. PMID 29290515
- [Result] Eschenbacher WL. Defining Airflow Obstruction. Chronic Obstr Pulm Dis. 2016;3(2):515-518. doi: 10.15326/jcopdf.3.2.2015.0166. PMID 27239557
- [Result] Galant SP, Komarow HD, Shin HW, Siddiqui S, Lipworth BJ. The case for impulse oscillometry in the management of asthma in children and adults. Ann Allergy Asthma Immunol. 2017 Jun;118(6):664-671. doi: 10.1016/j.anai.2017.04.009. PMID 28583260
- [Result] Postma DS, Brightling C, Baldi S, Van den Berge M, Fabbri LM, Gagnatelli A, Papi A, Van der Molen T, Rabe KF, Siddiqui S, Singh D, Nicolini G, Kraft M; ATLANTIS study group. Exploring the relevance and extent of small airways dysfunction in asthma (ATLANTIS): baseline data from a prospective cohort study. Lancet Respir Med. 2019 May;7(5):402-416. doi: 10.1016/S2213-2600(19)30049-9. Epub 2019 Mar 12. PMID 30876830
- [Result] Kuo CW, Liao XM, Huang YC, Chang HY, Shieh CC. Bronchoscopy-guided bronchial epithelium sampling as a tool for selecting the optimal biologic treatment in a patient with severe asthma: a case report. Allergy Asthma Clin Immunol. 2019 Nov 27;15:76. doi: 10.1186/s13223-019-0378-6. eCollection 2019. PMID 31798645
- [Result] Parulekar AD, Diamant Z, Hanania NA. Role of biologics targeting type 2 airway inflammation in asthma: what have we learned so far? Curr Opin Pulm Med. 2017 Jan;23(1):3-11. doi: 10.1097/MCP.0000000000000343. PMID 27820746
- [Result] Li Y, Wang W, Lv Z, Li Y, Chen Y, Huang K, Corrigan CJ, Ying S. Elevated Expression of IL-33 and TSLP in the Airways of Human Asthmatics In Vivo: A Potential Biomarker of Severe Refractory Disease. J Immunol. 2018 Apr 1;200(7):2253-2262. doi: 10.4049/jimmunol.1701455. Epub 2018 Feb 16. PMID 29453280
- [Result] Liu S, Verma M, Michalec L, Liu W, Sripada A, Rollins D, Good J, Ito Y, Chu H, Gorska MM, Martin RJ, Alam R. Steroid resistance of airway type 2 innate lymphoid cells from patients with severe asthma: The role of thymic stromal lymphopoietin. J Allergy Clin Immunol. 2018 Jan;141(1):257-268.e6. doi: 10.1016/j.jaci.2017.03.032. Epub 2017 Apr 20. PMID 28433687
- [Result] Specjalski K, Niedoszytko M. MicroRNAs: future biomarkers and targets of therapy in asthma? Curr Opin Pulm Med. 2020 May;26(3):285-292. doi: 10.1097/MCP.0000000000000673. PMID 32101904